CLINICAL TRIAL: NCT06001385
Title: A Phase II Study of Reduced Dose Post Transplantation Cyclophosphamide as GvHD Prophylaxis in Adult Patients With Hematologic Malignancies Receiving HLA-Mismatched Unrelated Donor Peripheral Blood Stem Cell Transplantation
Brief Title: HLA-Mismatched Unrelated Donor Peripheral Blood Stem Cell Transplantation With Reduced Dose Post Transplantation Cyclophosphamide GvHD Prophylaxis
Acronym: OPTIMIZE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMIZE
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Acute Leukemia; Myelodysplastic Syndromes; Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia; Myeloproliferative Neoplasm; Lymphoma; Chronic Myelomonocytic Leukemia; Pro-Lymphocytic Leukemia; Myelofibrosis
Keywords: Lymphoma; Leukemia; Hematologic Diseases; Myelodysplastic Syndromes; Preleukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia , Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Disorders; Bone Marrow Diseases; Precancerous Conditions; Leukemia, Lymphoid; Leukemia, B-Cell; Leukemia, Myeloid; Cyclophosphamide; Mesna; Tacrolimus; Busulfan; Fludarabine; Total Body Irradiation; Melphalan; Mycophenolate mofetil; Reduced Dose Cyclophosphamide; Immunosuppressive Agents; Immunologic Factors; Physiological Effects of Drugs; Hematopoietic Stem Cell Transplantation; Peripheral Blood Stem Cells; Unrelated Donors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Myeloproliferative Disorders; Lymphoma; Leukemia, Myelomonocytic, Chronic; Leukemia, Prolymphocytic; Primary Myelofibrosis; Leukemia; Hematologic Diseases; Preleukemia; Leukemia, B-Cell; Leukemia, Biphenotypic, Acute; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Bone Marrow Diseases; Precancerous Conditions; Leukemia, Lymphoid; Leukemia, Myeloid | interventions — Busulfan; fludarabine; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; Cyclophosphamide; Mesna; Tacrolimus; Mycophenolic Acid; Patient Reported Outcome Measures; Melphalan; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Regimen A (MAC: Busulfan and Fludarabine, PBSC HCT; Reduce Dose PTCy (Experimental): Patients Receive:
  Patients receive:
  Busulfan (≥ 9 mg/kg total dose) IV or PO on days -6 to -3 Fludarabine (150 mg/m2 total dose) IV on days -6 to -2
  Patients receive a peripheral blood stem cell (PBSC) graft infusion from a mismatched unrelated donor on Day 0.
  Patients receive a reduced dose of cyclophosphamide (25mg/kg per dose) on Day 3 and Day 4 post-transplant.
  First 20 patients with a 4-6/8 mismatched unrelated donor will receive an alternate dose of post-transplant cyclophosphamide of 37.5 mg/kg on Days 3 and Day 4 post-transplant.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT); Drug: Post-Transplant Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient Reported Outcomes
- Regimen B (MAC: Fludarabine and TBI, PBSC HCT; Reduce Dose PTCy (Experimental): Patients receive:
  Fludarabine (90 mg/m2 total dose) IV on days -7 to -5 Total body irradiation (TBI) (1200 cGy total dose) on days -4 to -1
  Patients receive a peripheral blood stem cell (PBSC) graft infusion from a mismatched unrelated donor on Day 0.
  Patients receive a reduced dose of cyclophosphamide (25mg/kg per dose) on Day 3 and Day 4 post-transplant.
  First 20 patients with a 4-6/8 mismatched unrelated donor will receive an alternate dose of post-transplant cyclophosphamide of 37.5 mg/kg on Days 3 and Day 4 post-transplant.
  Interventions: Drug: Fludarabine; Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT); Drug: Post-Transplant Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient Reported Outcomes; Radiation: Total-body irradiation
- Regimen C (RIC: Fludarabine and Busulfan; PBSCT HCT; Reduced Dose PTCy (Experimental): Patients receive:
  Fludarabine (150-180 mg/m2 total dose) IV on days -6 to -2 Busulfan (less than or equal to 8 mg/kg PO or 6.4 mg/kg IV) on days -5 and -4
  Patients receive a peripheral blood stem cell (PBSC) graft infusion from a mismatched unrelated donor on Day 0.
  Patients receive a reduced dose of cyclophosphamide (25mg/kg per dose) on Day 3 and Day 4 post-transplant.
  First 20 patients with a 4-6/8 mismatched unrelated donor will receive an alternate dose of post-transplant cyclophosphamide of 37.5 mg/kg on Days 3 and Day 4 post-transplant.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT); Drug: Post-Transplant Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient Reported Outcomes
- Regimen D (RIC: Fludarabine and Melphalan; PBSCT HCT; Reduced Dose PTCy (Experimental): Patients receive:
  Fludarabine (125-150 mg/m2 total dose) IV on days -7 to -3 Melphalan (100-140 mg/m2) IV on day -1
  Patients receive a PBSC graft infusion from a mismatched unrelated donor on Day 0.
  Patients receive a reduced dose of cyclophosphamide (25mg/kg per dose) on Day 3 and Day 4 post-transplant.
  First 20 patients with a 4-6/8 mismatched unrelated donor will receive an alternate dose of post-transplant cyclophosphamide of 37.5 mg/kg on Days 3 and Day 4 post-transplant.
  Interventions: Drug: Fludarabine; Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT); Drug: Post-Transplant Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient Reported Outcomes; Drug: Melphalan
- Regimen E (NMA: Fludarabine, Cyclophosphamide, and TBI; PBSCT HCT; Reduced Dose PTCy (Experimental): Patients receive:
  Fludarabine (150mg/m2 total dose) IV on days -6 to -2 Cyclophosphamide (29-50mg/kg) IV on days -6 and -5 TBI (200cGy) on day -1
  Patients receive a PBSC graft infusion from a mismatched unrelated donor on Day 0.
  Patients receive a reduced dose of cyclophosphamide (25mg/kg per dose) on Day 3 and Day 4 post-transplant.
  First 20 patients with a 4-6/8 mismatched unrelated donor will receive an alternate dose of post-transplant cyclophosphamide of 37.5 mg/kg on Days 3 and Day 4 post-transplant.
  Interventions: Drug: Fludarabine; Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT); Drug: Post-Transplant Cyclophosphamide; Drug: Mesna; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Other: Patient Reported Outcomes; Radiation: Total-body irradiation; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Busulfan — Given IV or PO pre-transplant as part of conditioning regimen
  Other Names: Busulfex®
  Arms: Regimen A (MAC: Busulfan and Fludarabine, PBSC HCT; Reduce Dose PTCy; Regimen C (RIC: Fludarabine and Busulfan; PBSCT HCT; Reduced Dose PTCy
Drug: Fludarabine — Given IV pre-transplant as part of conditioning regimen
  Other Names: Fludara®
Procedure: PBSC Hematopoietic Stem Cell Transplantation (HSCT) — Peripheral blood stem cell graft is infused from a mismatched unrelated donor on Day 0
  Other Names: PBSC HSCT; PBSC HCT; PBSC Transplantation; PBSCT
Drug: Post-Transplant Cyclophosphamide — Cyclophosphamide (25mg/kg) is administered on Day 3 and Day 4 post-transplant as an IV infusion over 1-2 hours.
  First 20 subjects with a 4-6/8 HLA mismatched unrelated donor will receive an intermediate dose of post-transplant cyclophosphamide of 37.5 mg/kg Day 3 and Day 4 post-transplant.
  Other Names: Cytoxan®; PTCy
Drug: Mesna — Mesna is given in divided doses IV 30 min pre- and at 3, 6, and 8 hours post cyclophosphamide.
  Other Names: Mesnex®
  Arms: Regimen E (NMA: Fludarabine, Cyclophosphamide, and TBI; PBSCT HCT; Reduced Dose PTCy
Drug: Tacrolimus — Tacrolimus is given at a dose of 0.05 mg/kg PO or an IV dose of 0.03 mg/kg of ideal body weight (IBW) starting on Day +5 post-transplant with taper recommended at Day + 90 and finished by Day +180.
Drug: Mycophenolate Mofetil — Mycophenolate mofetil (MMF) is given at a dose of 15 mg/kg three times daily IV or PO from Day +5 to Day +35 post-transplant.
  Other Names: MMF; Cellcept®
Other: Patient Reported Outcomes — Survey assessments will be administered to study participants pre transplant, at Day + 100, Day + 180, and Day +365 post transplant.
  Other Names: PRO
Drug: Melphalan — Given IV pre transplant as part of conditioning regimen
  Arms: Regimen D (RIC: Fludarabine and Melphalan; PBSCT HCT; Reduced Dose PTCy
Radiation: Total-body irradiation — Administered pre-transplant as part of conditioning regimen
  Other Names: TBI
  Arms: Regimen B (MAC: Fludarabine and TBI, PBSC HCT; Reduce Dose PTCy; Regimen E (NMA: Fludarabine, Cyclophosphamide, and TBI; PBSCT HCT; Reduced Dose PTCy
Drug: Cyclophosphamide — Given IV pre-transplant as part of conditioning regimen
  Other Names: Cytoxan®
  Arms: Regimen E (NMA: Fludarabine, Cyclophosphamide, and TBI; PBSCT HCT; Reduced Dose PTCy

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of Reduced Dose Post-Transplant Cyclophosphamide (PTCy) in patients with hematologic malignancies after receiving an HLA-Mismatched Unrelated Donor (MMUD) . The main question[s] it aims to answer are:

* Does a reduced dose of PTCy reduce the occurrence of infections in the first 100 days after transplant?
* Does a reduced dose of PTCy maintain the same level of protection against Graft Versus Host Disease (GvHD) as the standard dose of PTCy?

ELIGIBILITY:
Stratum 1 Recipient Inclusion Criteria:

1. Age ≥ 18 years and < 66 years (chemotherapy-based conditioning) or < 61 years (total body irradiation [TBI]-based conditioning) at the time of signing informed consent
2. Patient or legally authorized representative has the ability to provide informed consent according to the applicable regulatory and institutional requirements.
3. Stated willingness to comply with all study procedures and availability for the duration of the study.
4. Planned MAC regimen as defined per study protocol
5. Available partially HLA-MMUD (4/8-7/8 at HLA-A, -B, -C, and -DRB1 is required) with age ≥ 18 and ≤ 40 years (≤ 35 preferred).
6. Product planned for infusion is MMUD T-cell replete PBSC allograft
7. HCT-CI < 5. The presence of prior malignancy will not be used to calculate HCT-CI for this trial to allow for the inclusion of patients with secondary or therapy-related AML or MDS.
8. One of the following diagnoses:

   1. Acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), or other acute leukemia in 1st remission or beyond with ≤ 5% marrow blasts and no circulating blasts or evidence of extra-medullary disease. Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   2. Patients with MDS with no circulating blasts and with < 10% blasts in the bone marrow (higher blast percentage allowed in MDS due to lack of differences in outcomes with < 5% or 5-10% blasts in MDS). Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
9. Cardiac function: Left ventricular ejection fraction ≥ 45% based on most recent echocardiogram or multi-gated acquisition scan (MUGA) results.
10. Estimated creatinine clearance ≥ 45mL/min calculated by equation.
11. Pulmonary function: diffusing capacity of the lungs for carbon monoxide (DLCO) corrected for hemoglobin > 50% and forced expiratory volume in first second (FEV1) predicted > 50% based on most recent pulmonary function test (PFT) results
12. Liver function acceptable per local institutional guidelines
13. KPS of ≥ 70%

Stratum 2 Recipient Inclusion Criteria:

1. Age ≥18 years at the time of signing informed consent
2. Patient or legally authorized representative has the ability to provide informed consent according to the applicable regulatory and local institutional requirements.
3. Stated willingness to comply with all study procedures and availability for the duration of the study.
4. Planned NMA/RIC regimen per study protocol
5. Available partially HLA-MMUD (4/8-7/8 at HLA-A, -B, -C, and -DRB1 is required) with age ≥ 18 and ≤ 40 years (≤ 35 preferred).
6. Product planned for infusion is MMUD T-cell replete PBSC allograft
7. One of the following diagnoses:

   1. Patients with acute leukemia or chronic myeloid leukemia (CML) with no circulating blasts, no evidence of extramedullary disease, and with < 5% blasts in the bone marrow.

      Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   2. Patients with MDS with no circulating blasts and with < 10% blasts in the bone marrow (higher blast percentage allowed in MDS due to lack of differences in outcomes with < 5% or 5-10% blasts in MDS.) Documentation of bone marrow assessment will be accepted within 45 days prior to the anticipated start of conditioning.
   3. Patients with chronic lymphocytic leukemia (CLL) or other leukemias (including prolymphocytic leukemia) with chemosensitive disease at time of transplantation
   4. Higher risk CMML according to CMML-specific prognostic scoring system or high risk MDS/MPN not otherwise specified are eligible, provided there is no evidence of high-grade bone marrow fibrosis or massive splenomegaly at the time of enrollment.
   5. Patients with lymphoma with chemosensitive disease at the time of transplantation
8. Cardiac function: Left ventricular ejection fraction ≥ 40% based on most recent echocardiogram or MUGA results with no clinical evidence of heart failure
9. Estimated creatinine clearance ≥ 45mL/min calculated by equation
10. Pulmonary function: DLCO corrected for hemoglobin > 50% and FEV1 predicted >50% based on most recent PFT results
11. Liver function acceptable per local institutional guidelines
12. KPS of ≥ 60%

Stratum 3 Recipient Inclusion Criteria:

1. Age ≥18 years at the time of signing informed consent
2. Patient or legally authorized representative has the ability to provide informed consent according to the applicable regulatory and local institutional requirements.
3. Stated willingness to comply with all study procedures and availability for the duration of the study.
4. Planned NMA/RIC regimen per study protocol
5. Available partially HLA-MMUD (4/8-7/8 at HLA-A, -B, -C, and -DRB1 is required) with age ≥ 18 and ≤ 40 years (≤ 35 preferred).
6. Product planned for infusion is MMUD T-cell replete PBSC allograft
7. Diagnosis of primary myelofibrosis with risk features making them eligible for HCT. Myelofibrosis secondary to essential thrombocythemia, polycythemia vera, or MDS with grade 4 fibrosis are also eligible. Patients with a myelofibrosis diagnosis require sponsor approval before enrolling.
8. Cardiac function: Left ventricular ejection fraction ≥ 40% based on most recent echocardiogram or MUGA results with no clinical evidence of heart failure
9. Estimated creatinine clearance ≥ 45 mL/min calculated by equation
10. Pulmonary function: DLCO corrected for hemoglobin > 50% and FEV1 predicted >50% based on most recent PFT results
11. Liver function acceptable per local institutional guidelines
12. KPS of ≥ 60%

Donor Inclusion Criteria (note: donors are not research subjects):

1. Must be unrelated to the subject and high-resolution HLA-matched at 4/8, 5/8, 6/8, or 7/8 (HLA-A, -B, -C, and -DRB1.
2. Donor must be typed at high-resolution for a minimum of HLA-A, -B, -C, -DQB1, and -DPB1.
3. Age ≥ 18 years and ≤ 40 years at the time of signing informed consent for PBSC donation. Note: donors are preferred to be ≤ 35.
4. Meet the donor registries' medical suitability requirements for PBSC donation.
5. Must undergo eligibility screening according to current Food and Drug Administration (FDA) requirements. Donors who do not meet one or more of the donor screening requirements may donate under urgent medical need.
6. Must agree to donate PBSC.
7. Must have the ability to give informed consent according to standard (non-study) informed consent according to applicable donor regulatory requirements.

Recipient Exclusion Criteria (Strata 1, 2, and 3):

1. Suitable HLA-matched related or 8/8 high-resolution matched unrelated donor available
2. Subject unwilling or unable to give informed consent, or unable to comply with the protocol including required follow-up and testing
3. Subjects with a prior allogeneic transplant
4. Subjects with an autologous transplant within the past 3 months
5. Females who are breast-feeding or pregnant
6. Uncontrolled bacterial, viral, or fungal infection at the time of the transplant preparative regimen
7. Concurrent enrollment on a preventative GvHD and/or infectious disease prevention clinical trial.
8. Subjects who undergo desensitization to reduce anti-donor HLA antibody levels prior to transplant.
9. Patients who are HIV+ with persistently positive viral load. HIV-infected patients on effective anti-retroviral therapy (ART) with undetectable viral load within 6 months are eligible for this trial. Patients with well controlled HIV are eligible provided resistance panels are negative, the patient is compliant with ART, and their disease remains well controlled.

Donor Exclusion Criteria:

1. Donor unwilling or unable to donate.
2. Recipient positive for HLA antibodies against a mismatched HLA in the selected donor determined by the presence of donor specific HLA antibodies (DSA) to any mismatched HLA allele/antigen at any of the following loci (HLA-A, -B, -C, -DRB1, DRB3, DRB4, DRB5, -DQA1, - DQB1, -DPA1, -DPB1) with median fluorescence intensity (MFI) >3000 by microarray-based single antigen bead testing. In patients receiving red blood cell or platelet transfusions, DSA evaluation must be performed or repeated post-transfusion and prior to donor mobilization and initiation of recipient preparative regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Infection Free Survival | 100 days post-HCT
  Survival at 100 days without grades 2-3 infections (per BMT CTN grading criteria)

SECONDARY OUTCOMES:
Overall Survival | 1-year post-HCT
  Defined as time interval between date of transplant and death from any cause
Progression-free survival | 1-year post-HCT
  Defined as disease relapse or progression, or death by any cause
Infection-free survival | 1-year post-HCT
  Defined as death and grades II-III infection (per BMT CTN criteria)
Graft versus host disease relapse free survival | 1-year post-HCT
  Defined as relapse or progression of underling disease (by 1 year), grade III-IV acute GvHD (by 6 months), chronic GvHD requiring systemic immune suppression (by 1 year), or death by any cause (by 1 year).
Non-relapse mortality | 1-year post-HCT
  Defined as death without evidence of disease progression or recurrence
Cumulative incidence of neutrophil recovery | Day 28 post-HCT
  Defined as achieving an absolute neutrophil count (ANC) greater than or equal to 500/mm3 for three consecutive measurements on three different days
Cumulative incidence of platelet recovery | Day 28 post-HCT
  Defined as platelet count ≥20,000/mm^3 or ≥50,000/mm^3 with no platelet transfusions within seven days.
Cumulative incidence of primary and secondary graft failure | Day 28 and 1-year post-HCT
  Primary graft failure is defined as no neutrophil recovery to ≥ 500 cells/mm3 by Day 28 post HCT.
  Secondary graft failure is defined as as initial neutrophil count recovery followed by subsequent decline in absolute neutrophil counts <500 cells/mm3, unresponsive to growth factor therapy, but cannot be explained by infection, disease relapse, or medications.
Donor T-Cell Chimerism | Day 28, 100 and 365 post-HCT
  Defined as percent of donor chimerism via peripheral blood
Cumulative incidence of acute GvHD | Day 100 and Day 180 post-HCT
  Defined as cumulative incidence of grades II-IV acute GvHD
Cumulative incidence of chronic GvHD | 1-year post-HCT
Cumulative incidence of grade 2-3 bacterial, fungal, and viral infections | Day 100 and 1-year post-HCT
  Defined as grades 2-3 infection as defined by BMT CTN grading criteria.
Cumulative incidence of grades 2-3 BK virus hemorrhagic cystitis | 1-year post-HCT
  Defined as incidence of BK virus hemorrhagic cystitis per BMT CTN grading criteria
Cumulative incidence of relapse/progression | 1-year post-HCT
  Defined as disease relapse or progression from Day 0 to 1-year post-HCT
Overall Toxicity | 1-year post-HCT
  To tabulate adverse events (AEs, experienced by recipients, defined as grade 3-5 unexpected and grade 5 expected AEs according to CTCAE v5
Incidence and Severity of cytokine release syndrome | within 14 days post-HCT
  Defined and graded using the ASTCT grading criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Devine, MD, Principal Investigator — NMDP; Jeffery Auletta, MD, Study Chair — NMDP
Locations (32):
- United States (32):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Honor Health, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Colorado Blood Cancer Institute at Presbyterian St. Luke's, Denver, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Greenbaum Cancer Center University of Maryland, Baltimore, Maryland
  - Tufts University, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Barnes Jewish Hospital / Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center - Adults, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Center for Bone Marrow Transplantation at Geisinger, Danville, Pennsylvania
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - TriStar Centennial, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Methodist Hospital San Antonio, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No